CLINICAL TRIAL: NCT07120321
Title: Twelve-Month Prospective Evaluation of Clinical and Radiographic Outcomes of Pulpotomy Materials in Primary Molars
Brief Title: Pulpotomy Materials in Primary Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sacide Duman (Other)
Collaborators: Inonu University (Other)
Responsible Party: Sponsor-Investigator, Sacide Duman, Assoc. Prof. Dr., Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/77-INUDF; TSA-2021-2486. (Other Grant/Funding Number: Inonu University Scientific Research Projects Unit (BAP))
Record Dates: First submitted 2025-07-21; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries; Pulpitis
Keywords: Pulpotomy; Primary Molars; Calcium Silicate; Sodium Hypochlorite; Pediatric Dentistry; Vital Pulp Therapy
MeSH Terms: conditions — Dental Caries; Pulpitis | interventions — mineral trioxide aggregate; ProRoot MTA; tricalcium silicate; ferric sulfate

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical trial with a split-mouth design where each participant receives multiple interventions on different teeth.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors are blinded to the treatment allocation to reduce assessment bias. Participants, care providers, and investigators are aware of the assigned treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MTA Group (Experimental): Primary molars treated with Mineral Trioxide Aggregate (MTA) as the pulpotomy medicament.
  Interventions: Drug: Mineral Trioxide Aggregate (MTA)
- Biodentine Group (Experimental): Primary molars treated with Biodentine as the pulpotomy medicament.
  Interventions: Drug: Biodentine
- Ferric Sulfate Group (Experimental): Primary molars treated with 15.5% Ferric Sulfate as the pulpotomy medicament.
  Interventions: Drug: Ferric Sulfate
- Sodium Hypochlorite Gel Group (Experimental): Primary molars treated with 5% Sodium Hypochlorite gel as the pulpotomy medicament.
  Interventions: Drug: Sodium hypochlorite gel application

INTERVENTIONS:
Drug: Mineral Trioxide Aggregate (MTA) — Used as the capping agent after coronal pulp removal in primary molars.
  Other Names: MTA; ProRoot MTA
  Arms: MTA Group
Drug: Biodentine — Used as a bioactive pulpotomy agent following coronal pulp amputation.
  Other Names: Septodont Biodentine; Calcium Silicate Cement
  Arms: Biodentine Group
Drug: Ferric Sulfate — 15.5% Ferric Sulfate applied to pulp stumps for 15 seconds during pulpotomy procedure.
  Other Names: Astringedent; FS
  Arms: Ferric Sulfate Group
Drug: Sodium hypochlorite gel application — 5% NaOCl gel applied to pulp tissue during pulpotomy for its hemostatic and disinfectant effects.
  Other Names: NaOCl gel; Hypochlorite gel
  Arms: Sodium Hypochlorite Gel Group

SUMMARY:
This randomized clinical trial aims to compare four different materials used in a dental procedure called pulpotomy. Pulpotomy is commonly performed on primary molars (back teeth in children) to treat deep cavities and preserve the tooth. Children aged 4 to 7 who need this procedure will receive one of four materials: Mineral Trioxide Aggregate (MTA), Biodentine, Ferric Sulfate, or Sodium Hypochlorite gel. The treated teeth will be checked at 6 and 12 months to evaluate the success of each material. The goal is to identify the most effective and reliable material for pulpotomy in primary molars.

DETAILED DESCRIPTION:
Vital pulpotomy is a conservative and widely used treatment to maintain the function of primary molars affected by deep carious lesions. The choice of pulpotomy medicament plays a significant role in the long-term success of the procedure.

This randomized clinical trial is designed to compare the clinical and radiographic success rates of four pulpotomy agents: Mineral Trioxide Aggregate (MTA), Biodentine, Ferric Sulfate (FS), and Sodium Hypochlorite gel (NaOCl gel).

A total of 88 mandibular second primary molars in children aged 4 to 7 years will be included. After coronal pulp removal, one of the four materials will be applied to the pulp tissue. All treated teeth will be restored with stainless steel crowns. Follow-up evaluations will be performed at 6 and 12 months to assess the clinical and radiographic success of each material.

The findings from this study are expected to help determine the most effective and reliable pulpotomy material for use in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 4 and 7 years
* At least one primary molar indicated for pulpotomy
* No spontaneous pain or systemic infection
* Cooperative behavior according to the Frankl Behavior Rating Scale (scores 3 or 4)
* Signed informed consent from parents or legal guardians

Exclusion Criteria:

* Medically compromised children or presence of systemic diseases (e.g., bleeding disorders, immunodeficiency)
* Uncooperative behavior (Frankl rating 1 or 2)
* Primary teeth with signs of pulpal necrosis, abscess, sinus tract, or non-restorable crown
* History of allergy to any materials used in the study

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinical success after pulpotomy in primary molars | 12 months after pulpotomy
  Clinical success is defined as the absence of spontaneous pain, swelling, sinus tract, or abnormal mobility in the treated tooth during clinical examination.

SECONDARY OUTCOMES:
Number of participants with radiographic success after pulpotomy in primary molars | 12 months after pulpotomy
  Radiographic success is defined as the absence of internal/external root resorption, periapical or furcal radiolucency, and periodontal ligament widening.

CONTACTS AND LOCATIONS:
Overall Officials: sacide duman, Assoc Prof, Principal Investigator — Inonu University, Faculty of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Inonu University, Faculty of Dentistry, Department of Pediatric Dentistry, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This study does not plan to share individual participant data due to privacy concerns and institutional data protection policies. Data may be available upon reasonable request and with appropriate ethical approvals.

REFERENCES:
- [Derived] Vural H, Senem Ozsunkar P, Duman S, Syed AZ, Tirasci G. Clinical and radiographic outcomes of four pulpotomy agents in primary molars: a prospective randomized controlled trial. Odontology. 2025 Dec 7. doi: 10.1007/s10266-025-01281-4. Online ahead of print. PMID 41353690

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT07120321/Prot_SAP_000.pdf